CLINICAL TRIAL: NCT05832684
Title: A Phase I/II Clinical Study to Evaluate the Safety and Efficacy of ZVS101e Administered as a Single Monocular Subretinal Injection in Subjects With Bietti's Crystalline Dystrophy (BCD)
Brief Title: Safety and Efficacy of ZVS101e in Patients With Bietti 's Crystalline Dystrophy
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chigenovo Co., Ltd (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZYA-2022-001
Record Dates: First submitted 2023-04-02; First posted 2023-04-27 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Bietti's Crystalline Dystrophy
MeSH Terms: conditions — Bietti Crystalline Dystrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Dose escalation and expansion of ZVS101e. All patients enrolled in the study will receive a single subretinal injection of ZVS101e in one eye.
  Interventions: Drug: ZVS101e

INTERVENTIONS:
Drug: ZVS101e — ZVS101e contains recombinant adeno-associated virus serotype 8 (rAAV8) vectors which carry human wild type CYP4V2 gene.
  Other Names: rAAV2/8-hCYP4V2; rAAV8-hCYP4V2; AAV8-hCYP4V2

SUMMARY:
The purpose of this study was to evaluate the safety and efficacy of ZVS101e administered by subretinal injection in subjects with Bietti's crystalline dystrophy (BCD) and to select the optimal effective dose.

DETAILED DESCRIPTION:
This is a single-arm, open-label, and multi-center study of ZVS101e in patients with BCD. Up to 24 subjects are expected to be enrolled. Each participant will receive ZVS101e by subretinal injection in one eye on a single occasion. Safety, efficacy and vector shedding characteristics of ZVS101e are then measured over 180 days. Participants will subsequently enter a long-term follow-up study over a 4.5-year period.

ELIGIBILITY:
Inclusion Criteria:

* 1. Fully understand the purpose and requirements of this trial, voluntarily participate in the clinical trial, sign the informed consent form, and be able to complete the whole trial processes as required by the protocol;
* 2. Patients with clinical diagnosis of Bietti's crystalline dystrophy (BCD) (age ≥ 18 years) (including the critical value, and the age is based on the time of signing the informed consent form);
* 3. Genetic test confirmed to carry two pathogenic variants of CYP4V2 and carry no pathogenic mutations of other ophthalmic genetic diseases;
* 4. The study eye must meet the following requirements: Best-corrected visual acuity between 2.3 LogMAR and 0.5 LogMAR (including 2.3 LogMAR and 0.5 LogMAR).

Exclusion Criteria:

* 1. Subjects with insufficient viable retinal cells, or macular retinal less than 100 μm thick;
* 2. Pre-existing eye conditions in the study eye that the investigator determines could interfere with ocular evaluation, preclude surgery, interfere with interpretation of study endpoints or pose surgical complications;
* 3. The study eye has been treated with the following intraocular procedures: retinal detachment surgery, vitrectomy;
* 4. The study eye has been treated with other drugs within 3 months that could affect the evaluation of the investigational drug (such as ranibizumab, bevacizumab, aflibercept, conbercept);
* 5. Currently taking or may require systemic medications that can cause ocular toxicity, such as psoralen, risedronate, or tamoxifen;
* 6. Those with the following laboratory abnormalities which are clinically significant:

  * Liver function: chronic liver disease, ALT increased > 2 times the upper limit of normal;
  * Hypertension, mean SBP ≥ 160 mmHg or mean DBP ≥ 100 mmHg;
  * Coagulation function (prothrombin time ≥ upper limit of normal (3 seconds' longer), activated partial thromboplastin time ≥ upper limit of normal (10 seconds' longer));
  * Serum virology test: Active hepatitis B, hepatitis C virus antibody (HCV-Ab), human immunodeficiency virus antibody (HIV-Ab) or syphilis antibody positive;
* 7. Patients with rAAV8 neutralizing antibody titer ≥ 1:1000;
* 8. Complicating systemic diseases (such as medical conditions causing immunosuppression) that would preclude the gene transfer, ocular surgery and drug in vivo activity;
* 9. Known drug allergy to the drug planned to be used in the study;
* 10. Patients who cannot communicate or cooperate with medical staff due to neurological, mental illness or language disorder, which affects patient compliance;
* 11. Treatment of either eye with gene therapy drugs for BCD and other ocular diseases, including but not limited to other viral vector gene therapies, mRNA therapy, etc.;
* 12. Has or has had a systemic immune-compromising disease;
* 13. Subjects of reproductive age without any effective contraception and female subjects who have tested positive for pregnancy or are lactating at screening or baseline;
* 14. A condition that, in the opinion of the investigator, would preclude participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-02-20 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of ocular and systemic adverse events (AEs) after ZVS101e treatment | Up to day 180
  An adverse event (AE) is any untoward medical occurrence in a clinical investigation participant administered a product; the event will not need to have a causal relationship with the treatment.
Incidence of ocular and systemic serious adverse events (SAEs) after ZVS101e treatment | Up to day 180
  A serious adverse event (SAE) is any untoward medical occurrence at any dose that leading to the following:
  Results in death; Life-threatening, refers to an event in which the patient is at risk of death at the time of the event; it does not refer to an event which hypothetically might have caused death if it were more severe; Significant or permanent disability/incapacity, where disability refers to a serious disruption and damage of a person's ability to perform normal life functions; Requires inpatient hospitalization or prolongation of existing hospitalization; Congenital anomaly or birth defect; Other medically important events.
Mean change from baseline in BCVA (LogMAR) | Up to day 180
  BCVA of both eyes will be assessed using the early treatment of diabetic retinopathy study (ETDRS) chart.

SECONDARY OUTCOMES:
Change from Baseline in visual field | Up to day 180
  Visual field will be assessed by Humphrey perimetry, changes in retinal light sensitivity will be analyzed.
Change from Baseline in contrast sensitivity | Up to day 180
  Change from baseline in contrast sensitivity at all spatial frequency will be measured using the CSV-1000E instrument.
Change from Baseline in microperimetry | Up to day 180
  Microperimetry will be measured using MP-3，changes in retinal sensitivity (dB) will be analyzed.
Change from Baseline in mfERG | Up to day 180
  The measurement will be performed based on the standards of international society for clinical electrophysiology of vision (ISCEV). Response Amplitude Density will be analyzed.
Change from Baseline in retinal thickness | Up to day 180
  Retinal thickness will be assessed for both eyes using OCT.
Change from Baseline in NEI VFQ-25 total score | Up to day 180
  National eye institute 25-item visual function questionnaire (NEI VFQ-25) consists of a base set of 25 vision-targeted questions representing 11 vision-related constructs. All items are scored so that a high score represents better functioning. Each item is then converted to a 0 to 100 scale so that the lowest and highest possible scores are set at 0 and 100 points, respectively.
Change from Baseline in color vision | Up to day 180
  Subjects' color vision was classified and graded by having them identify the pictures within Color Vision Examination Plates.

OTHER OUTCOMES:
Change from Baseline in multi-luminance mobility test (MLMT) | Up to day 180
  MLMT was assessed using both eyes at 1 or more of 7 levels of illumination, ranging from 400 lux (a brightly lit office) to 1 lux (a moonless summer night).

CONTACTS AND LOCATIONS:
Overall Officials: Xiaorong Li, MD, Principal Investigator — Tianjin Medical University Eye Hospital
Locations (3):
- China (3):
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Tianjin Medical University Eye Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jia R, Meng X, Chen S, Zhang F, Du J, Liu X, Yang L. AAV-mediated gene-replacement therapy restores viability of BCD patient iPSC derived RPE cells and vision of Cyp4v3 knockout mice. Hum Mol Genet. 2023 Jan 1;32(1):122-138. doi: 10.1093/hmg/ddac181. PMID 35925866
- [Background] Wang J, Zhang J, Yu S, Li H, Chen S, Luo J, Wang H, Guan Y, Zhang H, Yin S, Wang H, Li H, Liu J, Zhu J, Yang Q, Sha Y, Zhang C, Yang Y, Yang X, Zhang X, Zhao X, Wang L, Yang L, Wei W. Gene replacement therapy in Bietti crystalline corneoretinal dystrophy: an open-label, single-arm, exploratory trial. Signal Transduct Target Ther. 2024 Apr 24;9(1):95. doi: 10.1038/s41392-024-01806-3. PMID 38653979